CLINICAL TRIAL: NCT01588132
Title: First Assessment of the Glycoprotein Ib-IV-V Complex Antagonist Anfibatide in Healthy Human Volunteers
Brief Title: Anfibatide Phase 1 Clinical Trial in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Principal Investigator, Vivian Fung, Ph.D, Lee's Pharmaceutical Limited
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: LeesPharm_Anfibatide_Phase1
Record Dates: First submitted 2012-04-25; First posted 2012-04-30 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Heart Disease; Coagulation Disorder
MeSH Terms: conditions — Coronary Disease; Hemostatic Disorders | interventions — agkisacucetin protein, Agkistrodon acutus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (11):
- Single dose gourp 1 (Experimental): Anfibatide injection at the concentration of 0.33μg/60kg in healthy volunteers
  Interventions: Drug: Anfibatide
- Single dose group 2 (Experimental): Anfibatide injection at the concentration of 0.66μg/60kg in healthy volunteers
  Interventions: Drug: Anfibatide
- Single dose groups 3 (Experimental): Anfibatide injection at the concentration of1.0μg/60kg in healthy volunteers
  Interventions: Drug: Anfibatide
- Single dose group 4 (Experimental): Anfibatide injection at the concentration of 1.5μg/60kg in healthy volunteers
  Interventions: Drug: Anfibatide
- Single dose group 5 (Experimental): Anfibatide injection at the concentration of 2.0μg/60kg in healthy volunteers
  Interventions: Drug: Anfibatide
- Single dose group 6 (Experimental): Anfibatide injection at the concentration of 3.0μg/60kg in healthy volunteers
  Interventions: Drug: Anfibatide
- Single dose group 7 (Experimental): Anfibatide injection at the concentration of 4.0μg/60kg in healthy volunteers
  Interventions: Drug: Anfibatide
- Single dose group 8 (Experimental): Anfibatide injection at the concentration of 5.0μg/60kg in healthy volunteers
  Interventions: Drug: Anfibatide
- Multiple dose group 9 (Experimental): Give intravenous injection of 3μg as the first dose and after 1.5 hours, infusion of the study product 0.12μg/h for 24 hours
  Interventions: Drug: Anfibatide
- Multiple dose group 10 (Experimental): Give intravenous injection of 3μg as the first dose and immediately infusion of the study product 0.12μg/h for 24 hours.
  Interventions: Drug: Anfibatide
- Multiple dose group 11 (Experimental): Give intravenous injection of 5μg as the first dose and immediately infusion of the study product 0.12μg/h for 24 hours
  Interventions: Drug: Anfibatide

INTERVENTIONS:
Drug: Anfibatide — 1. To investigate the safety and tolerability of single intravenous dose of Antiplatelet Thrombolysin for Injection of 0.33,0.66,1.0,1.5,2.0,3.0,4.0,5.0μg (body weight 60kg) in healthy volunteers.
  2. To investigate the safety and tolerability of continuous administration of three dose regimen: ① give intravenous injection of 3μg as the first dose and after 1.5 hours, infusion of the study product 0.12μg/h for 24 hours. ② give intravenous injection of 3μg as the first dose and immediately infusion of the study product 0.12μg/h for 24 hours. ③ give intravenous injection of 5μg as the first dose and immediately infusion of the study product 0.12μg/h for 24 hours.

SUMMARY:
In this 94 healthy subjects Phase I clinical trial, we assess the clinical profile of Anfibatide, a specific glycoprotein Ib antagonist. This study represents the first clinical evidence that Anfibatide exhibits strong anti-platelet effects, excellent reversibility, and low bleeding potential in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1) Healthy volunteers, aged 18-28 years, male and female were included, age difference less than 10 years;
* 2) Body weight: with body mass index (BMI) between 19-24, difference less than 10kg in the same group, BMI=body weight(kg)/height2;
* 3) Past medical history: no history of heart, liver, kidney, digestive tract, nervous system and metabolic disorder, or ulcer, significant hemorrhage, without the history of drug allergy and postural hypotension;
* 4) Medical examinations: with normal results in overall examinations (including heart rate, blood pressure, auscultation of heart and lung, palpation of liver and spleen, hepatic and renal function, hematology, coagulation function, urine analysis, stool analysis and occult blood test, electrocardiogram);
* 5) Have not received any medications within 2 weeks before the study;
* 6) Willing to participate in the study and give a signed informed consent form after understanding the study procedures and potential adverse reactions of the study product.

Exclusion Criteria:

* 1) History of HBV or HCV infection;
* 2) Addicted to smoking or alcohol;
* 3) Women during pregnancy, lactation or menstrual period;
* 4) Past history of hemoptysis, bloody stool, bleeding spots in the skin and mucous membrane, or hemorrhagic tendency (find themselves prone to bleeding in gums, nose, skin and mucous membrane, or hemoptysis);
* 5) History of active bleeding (such as peptic ulcer, hemorrhoids, active tuberculosis, subacute bacterial endocarditis, etc);
* 6) Blood platelet count less than 150×109;
* 7) Trauma history (e.g., craniocerebral trauma) recently;
* 8) Past history of unexplained syncope or convulsion;
* 9) History of organic or psychogenic disease or the disabled;
* 10) Persons who were unlikely to participate in the study (such as the infirm) in the investigator's opinion;
* 11) Have donated blood or experienced blood collection in other trials within 3 months.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety endpoints | 24 Hours
  To investigate the number of adverse events in patients with single or multiple intravenous injection/infusion of Antiplatelet

SECONDARY OUTCOMES:
Area Under Curve (AUC) | Predose, 0,1,2,3,4,6,8,12,24,48,72,96 Hours
  To observe area under curve characteristics of Anfibatide in single or multiple dose groups

REFERENCES:
- [Derived] Li BX, Dai X, Xu XR, Adili R, Neves MAD, Lei X, Shen C, Zhu G, Wang Y, Zhou H, Hou Y, Ni T, Pasman Y, Yang Z, Qian F, Zhao Y, Gao Y, Liu J, Teng M, Marshall AH, Cerenzia EG, Li ML, Ni H. In vitro assessment and phase I randomized clinical trial of anfibatide a snake venom derived anti-thrombotic agent targeting human platelet GPIbalpha. Sci Rep. 2021 Jun 3;11(1):11663. doi: 10.1038/s41598-021-91165-8. PMID 34083615